CLINICAL TRIAL: NCT02738723
Title: Stereotactic Body Radiation Therapy Compared With Intensity Modulated Radiation Therapy Concurrently With Chemotherapy in Treating Patients With Limited-Stage Small Cell Lung Cancer
Brief Title: SBRT Compared With IMRT Concurrently With Chemotherapy in Treating Patients With LS-SCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Xueqin Yang, Prof., Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STIM
Record Dates: First submitted 2016-03-25; First posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Small Cell Lung Cancer
Keywords: Limited-stage small cell lung cancer; Stereotactic body radiation therapy; Intensity modulated radiation therapy; Radiation; Chemotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GROUP 1 (Experimental): SBRT plus EP
  Interventions: Radiation: SBRT; Drug: EP
- GROUP 2 (Active Comparator): IMRT plus EP
  Interventions: Radiation: IMRT; Drug: EP

INTERVENTIONS:
Radiation: SBRT — 40 Gy for each patient. Patients receiving once-daily therapy ,4 Gy daily in 10 treatments over a period of two weeks.
  Arms: GROUP 1
Radiation: IMRT — 45 Gy for each patient，Accelerated twice-daily thoracic radiotherapy involved the administration of 1.5 Gy in 30 treatments over a period of three weeks.
  Arms: GROUP 2
Drug: EP — Etoposide 75mg/m2/iv over 90min through day 1 to day 4 and cisplatin 25mg/m2/iv over 30min through day 1 to day 3, repeat Q 3weeks. Continuous administration to six cycles or to disease progression, unacceptable toxicity or patients' refusal.

SUMMARY:
As stereotactic radiotherapy (SBRT) has been widely used in clinical practice at present, the aim of this study is to evaluate the efficacy and safety of stereotactic body radiation therapy compared with intensity modulated radiation therapy (IMRT) concurrently with EP regimen(cisplatin plus etoposide) in treating patients with limited-stage small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of SCLC
* limited-stage disease is defined as disease confined to the ipsilateral hemithorax, which can be safely encompassed within a radiation field
* No prior chemotherapy, or radiotherapy
* Performance status of 0, 1, 2 on the ECOG criteria.
* At least one unidimensional measurable lesion meeting Response Evaluation Criteria in Solid Tumors (RECIST. 2000).
* Adequate hematologic (neutrophil count >= 1,500/uL, platelets >= 100,000/uL), hepatic (transaminase =< upper normal limit(UNL)x2.5, bilirubin level =< UNLx1.5), and renal (creatinine =< UNL) function
* If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (intrauterine device [IUD], birth control pills, or barrier device) during and for 3 months after trial. If male, use of an approved contraceptive method during the study and 3 months afterwards. Females with childbearing potential must have a urine negative HCG test within 7 days prior to the study enrollment.

Exclusion Criteria:

* Non small cell lung cancer and carcinoid
* Supraclavicular lymphadenopathy
* Inability to comply with protocol or study procedures.
* Moderate and severe ventilation dysfunction
* Medically uncontrolled serious heart, lung, neurological, psychological, metabolic disease
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Pregnant or breast-feeding.
* Enrollment in other study within 30 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first，assessed up to 3 years

SECONDARY OUTCOMES:
Overall survival | From date of randomization until last survival confirm date or date of death from any cause, whichever came first, assessed up to 3 years
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | the first date of treatment to 3 months after the last dose of study drug
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Tumor response rate | the ratio between the number of responders and number of patients assessable for tumor response，assessed up to 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Xueqin Yang, PHD, Principal Investigator — Daping Hospital, Third Military Medical University
Locations (1):
- Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li C, Xiong Y, Zhou Z, Peng Y, Huang H, Xu M, Kang H, Peng B, Wang D, Yang X. Stereotactic body radiotherapy with concurrent chemotherapy extends survival of patients with limited stage small cell lung cancer: a single-center prospective phase II study. Med Oncol. 2014 Dec;31(12):369. doi: 10.1007/s12032-014-0369-x. Epub 2014 Nov 22. PMID 25416052
- [Background] Turrisi AT 3rd, Kim K, Blum R, Sause WT, Livingston RB, Komaki R, Wagner H, Aisner S, Johnson DH. Twice-daily compared with once-daily thoracic radiotherapy in limited small-cell lung cancer treated concurrently with cisplatin and etoposide. N Engl J Med. 1999 Jan 28;340(4):265-71. doi: 10.1056/NEJM199901283400403. PMID 9920950